CLINICAL TRIAL: NCT05565131
Title: Performance Measurement and Safety Evaluation of the PYTHEAS® ODYSSEE Angular Assistance System for Intra-pedicular Screw Placement in Adult Spine Surgery. First-in-human Study
Brief Title: Performance Measurement and Safety Evaluation of the PYTHEAS® ODYSSEE Angular Assistance System for Intra-pedicular Screw Placement in Adult Spine Surgery
Acronym: ODYSSEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IDIL/2021/VH-01
Record Dates: First submitted 2022-09-27; First posted 2022-10-04 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2022-09

CONDITIONS: Pedicle Screw; Surgical Navigation Systems
Keywords: Spinal deformity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PAtients requiring pedicle screw implantation (Experimental)
  Interventions: Device: Guided placement with PYTHEAS® ODYSSEE

INTERVENTIONS:
Device: Guided placement with PYTHEAS® ODYSSEE — Pre-surgery, the surgeon generates a 3D model of the spine from a preoperative CT scan During the perforation and insertion of the implant, the system indicates the orientation of the pedicle path and the current orientation of the instruments (perforation tool) with the orientation sensor (inertial sensor). The system also displays the position of the entry point of the planned pedicle path on the views.

SUMMARY:
Pedicle screw malposition is a common problem for spine surgeons. A poorly placed screw can lead to potentially serious complications (hemorrhage, paralysis) in the short- or medium-term. Accurate images during surgery facilitates preoperative planning and aids the placement of pedicle screws.

Surgical navigation covers all techniques and equipment (hardware and software) needed to perform a computer-assisted procedure with 3D image visualization of the surgical act.

Surgical navigation systems have been on the market for about 15 years. Surgical navigation increases the accuracy of pedicle screw placement. Many technologies are available, but they are expensive and often require extensive instrumentation.

The PYTHEAS® ODYSSEE angular assistance system has many advantages over more widely used systems. Indeed, this system provides surgeons with the necessary information to correctly insert pedicle screws during posterior spondylodesis procedures for the treatment of deformity, osteoarthritis (degenerative spine) and trauma.

Compared to competing solutions, the purpose of this device is to reduce pedicle screw malpositioning while offering minimal radiation exposure and the least possible impact on the conventional surgical workflow. It is a lightweight, efficient and easy-to-use medical device with 2-step functionality: 1) Surgical planning of pedicle screws based on a preoperative scan; 2) Angular assistance tool during surgery.

The study investigators wish to evaluate the performance and safety of the PYTHEAS® ODYSSEE medical device (not CE marked) as well as its usability in a pilot study of first use in humans.

Without a navigation system, the literature reports that on average 9 to 10% of perforations are incorrectly positioned by the "free hand" method. With the PYTHEAS® ODYSSEE angular assistance device, the study hypothesis is that this rate will be 5%, i.e. a 50% improvement.

ELIGIBILITY:
Inclusion Criteria:

* Patient with indication for posterior arthrodesis of at least 2 lumbar or thoracic vertebrae with placement of pedicle screws at vertebral level for :

  * Traumatology: fracture with significant vertebral compression or major kyphosis deformity, ligament and/or disc injury resulting in instability, with the need to free the marrow or nerve roots, OR
  * Deformity: idiopathic scoliosis with surgical indication for increased curvature, thoracic curvature greater than 45° or lumbar curvature greater than 35°, OR
  * Revision surgery for extension of the assembly in the presence of a possible adjacent syndrome responsible for instability and/or central or foraminal stenosis, OR
  * Degenerative: symptomatic spondylolisthesis, degenerative scoliotic deformity, narrow lumbar canal with canal release leading to instability, syndrome adjacent to a previously performed montage.
* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* Patients with contraindication to screw placement
* Patients with contraindication to CT scan
* Silicon allergy
* The subject is participating in a category 1 interventional study, or is in a period of exclusion determined by a previous study
* The patient is unable to express their consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Pregnant, parturient or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Accuracy of the PYTHEAS® ODYSSEE angular assistance device for directing the pedicle | Day 0
  Number of perforations with the correct direction/Total number of perforations performed. The correct direction will be determined using a palpator guide before screw placement, and considered satisfactory when the internal, external, superior and inferior walls of the intra-pedicular path are respected

SECONDARY OUTCOMES:
Correct screw positioning rate | Day 0
  Number of correctly positioned screws (in trans-pedicular) / Number of screws placed. Correct placement determined by CT scan performed immediately postoperatively
Adverse events | Day 0
  No adverse events are anticipated directly linked to the device
Operating time according to the calibration mode performed (specific mode/global mode) | Day 0
  Operating time (minutes): time from incision until closing indicated on the management software.
Surgeon's satisfaction with the calibration (specific/global) | Day 0
  5-level Likert scale + one item with open-ended. The questions asked will be:
  * Are you satisfied with the specific calibration?
  * Are you satisfied with the overall calibration?
  * What type of calibration would you prefer to use in practice? In which cases?
Surgeon's satisfaction with technical quality of the transfer between the PYTHEAS tablet and the computer for each procedure | Day 0
  5-level Likert scale + one item with open-ended. The questions asked will be:
  * Are you satisfied with the transfer time between the tablet and the computer?
  * Are you satisfied with the ease of transfer between the tablet and the computer?
Surgeon's satisfaction with tablet interaction | Day 0
  5-level Likert scale + suggestions for improvement. The questions asked will be:
  * Are you satisfied with the responsiveness of the tablet?
  * Are you satisfied with the interactivity of the tablet?
  * Are you satisfied with the quality of the images displayed by the tablet?
  * Suggestions for improvement.
Surgeon's reported overall usability of the PYTHEAS® ODYSSEE | Day 0
  The System Usability Scale (SUS): a 10-item questionnaire where a score of 75 or more is generally considered "good", and 50 to 75 is considered "fair" or "adequate". A score below 50 indicates major problems in terms of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Haignere, Principal Investigator — CHU de Nimes
Locations (2):
- France (2):
  - Hôpital Saint Joseph, Marseille
  - CHU de Nimes, Nîmes